CLINICAL TRIAL: NCT07322627
Title: ALDH2 Single Nucleotide Polymorphisms and Prognosis of Esophageal Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202511005RINA
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
Keywords: ALDH2; prognosis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study will use the remaining buffy coat frozen at -80°C, separated from whole blood, drawn from the subjects before cancer treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alcohol consumption, smoking, and betel nut chewing have been proven to be closely associated with the risk of esophageal cancer (EC). Recent studies have shown that alcohol-related detoxification genes in the ALDH family influence individual susceptibility to esophageal cancer. Aldehyde dehydrogenase 2 (ALDH2) is one of the most important enzymes in the ALDH family, involved in the metabolism of alcohol, acetaldehyde, and environmental aldehydes in the human body. We hypothesize that functional variations in ALDH2 may have a significant impact on the survival of esophageal cancer patients. This study aims to investigate the correlation between ALDH2 gene polymorphism and the survival of esophageal cancer patients.

DETAILED DESCRIPTION:
Many single nucleotide polymorphisms in genes involved in cell cycle progression, DNA repair, metabolism, and immune response have been implicated in susceptibility to cancers via different mechanisms, and thus might be used as diagnostic or prognostic markers of cancers. The most widely studied SNP for ALDH2 is rs671. Single nucleotide polymorphism of rs671 has two subtypes indicated as ALDH2*1 (G) and ALDH2*2 (A). The aldehyde dehydrogenase generated by ALDH2*2 (A) allele has a missense amino acid substitution (Glu504Lys in full length of cytoplasmic protein or Glu487Lys in mature mitochondrial protein) which causes low activity of ALDH2 in catalyzing the oxidation of toxic acetaldehyde into non-toxic acetic acid, leading to accumulation of acetaldehyde and increased incidence of cancers.

Around 40% of population in China carried the ALDH2*2 (A) allele; therefore, Chinese alcohol consumers with dysfunctional allele were more susceptible to upper aerodigestive tract cancers. A synergistic interaction between rs671 and alcohol consumption was also reported to increase the risk of head and neck cancer (HNC) and esophageal cancer by different research groups. Yokoyama et al. first found that Japanese male drinkers with inactivated ALDH2 were susceptible to multiple primary cancers with EC or oropharyngolaryngeal squamous cell carcinoma. Our previous study also demonstrated that ALDH2 rs671 was significantly associated with multiple primary cancers involving EC and head and neck cancer (HNC). However, ALDH2*2 (A) has also been reported to be a protective factor of colorectal cancer in a meta-analysis, and be indirectly associated with low risk of colorectal cancer, hepatocellular carcinoma, as well as digestive tract cancers among moderate alcohol consumers. Those with the ALDH2*2 variant often consumed less alcohol due to the acetaldehyde-induced unpleasant effects, which may decrease their risk for alcohol induced disorders. In addition, ALDH2*2 (A) was also reported to confer protective effect on ovarian cancer which was not related to alcohol consumption. To date, there were limited studies investigating the prognostic impact of ALDH2 SNPs on EC. In this study we aim to clarify the prognostic meanings of ALDH2 SNPs on EC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been pathologically confirmed to have esophageal cancer and who have previously signed consent forms indicating their willingness to provide remaining samples for subsequent studies.

Exclusion Criteria:

* Female patients or patients younger than 18 years old

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Totally up to 778 subjects with esophageal cancer will be retrospectively enrolled in National Taiwan University Hospital (NTUH) during the periods of study (from Dec 15, 2011 to Dec 31, 2024) with approval from the ethical committee of NTUH (202511005RINA).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
death | from the date of first diagnosis or undergoing esophagectomy to the end of 2024
  We will trace the patients with esophageal cancer for up to 150 months since the date of first diagnosis or undergoing esophagectomy, regarding their survival status. We will calculate the overall survival time (months) of each subject, and draw the overall survival curves for all patients based on their genotypes of SNP at ALDH2 locus.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan